CLINICAL TRIAL: NCT00209586
Title: A Phase III, Randomized, Open-label Study to Assess the Safety and Efficacy of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Patients Undergoing Flexible Bronchoscopy Procedures
Brief Title: A Study of AQUAVAN® Injection for Sedation in Elderly Patients Undergoing Flexible Bronchoscopy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient enrollment was stopped prior to completion of the study in order to re-evaluate the dosing regimen.
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Covance (Industry); Quest Pharmaceutical Services (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0409
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2012-01

CONDITIONS: Flexible Bronchoscopy
Keywords: Bronchoscopy; Sedation
MeSH Terms: interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
This study was designed to demonstrate that AQUAVAN® is effective in providing adequate sedation in patients undergoing flexible bronchoscopy as well as to assess the safety profile of AQUAVAN versus that of midazolam. Prior to the procedure, patients receive fentanyl citrate for pain management followed five minutes later by either AQUAVAN® Injection or midazolam HCl for sedation. During the procedure, study personnel assess the patient's vital signs and depth of sedation. After the procedure, the patient, physician, and an evaluator are asked to complete satisfaction surveys.

DETAILED DESCRIPTION:
This is a randomized, open-label study designed to assess the safety and efficacy of AQUAVAN® Injection versus midazolam HCl following pretreatment with an analgesic, fentanyl citrate injection, in producing sedation in patients undergoing a flexible bronchoscopy procedure. Randomization will be stratified by site. Following completion of pre-procedure sedation assessments, patients will be randomly assigned to 1 of the 2 i.v. treatment groups at a 3:1 (AQUAVAN® Injection: midazolam HCl) allocation ratio.

All study patients, irrespective of treatment group assignment, will receive fentanyl citrate injection as an analgesic pretreatment. Supplemental doses of fentanyl citrate injection may be administered if the patient reports pain or if inadequate analgesia is present as demonstrated by increased heart rate and/or blood pressure in the presence of adequate sedation. At no time should fentanyl citrate injection be administered to increase sedation levels. AQUAVAN® Injection and midazolam HCl will be administered to induce a state of adequate sedation, defined as a Modified Observer's Assessment of Alertness / Sedation (OAA/S) score of 4 or less. Supplemental doses will be administered to increase depth or duration of sedation. Supplemental doses will not be administered if the Modified OAA/S score is 2 or less or if there is no purposeful response to stimulation. The depth of sedation will be measured by the Modified OAA/S scale, a validated measure. Patient and Investigator assessments will be used to confirm that the depth of sedation provided met the goals of sedation, reduction of anxiety and reduced awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provided signed/dated Informed Consent and HIPAA Authorization after receiving a full explanation of the extent and nature of the study.
2. Patient was at least 18 years of age at the time of screening.
3. Female patient must have been surgically sterile, postmenopausal, or not pregnant or lactating, and must have been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predosing periods.
4. Patient met the American Society of Anesthesiologists (ASA) Physical Status Classification of I to III.

Exclusion Criteria:

1. Patient had a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic or benzodiazepine.
2. Patient did not meet nils per os (NPO) status per ASA Guideline or institution's guideline.
3. Patient had condition(s) that, in the opinion of the Investigator, could interfere with appropriate airway management.
4. Patient required artificial ventilation prior to the initiation of bronchoscopy or was admitted to the intensive care unit.
5. Patient had a history of mental or visual impairment that would not permit successful measurement of cognitive evaluations.
6. Patient was unwilling to adhere to pre- and postprocedural instructions.
7. The use of fentanyl or midazolam was contraindicated for the patient.
8. Patient had participated in an investigational study within 1 month prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Sedation success defined for a patient as having 3 consecutive Modified OAA/S scores <=4 and completing the procedure without requiring alternative sedative medications and without requiring manual or mechanical ventilation.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints
Time to Fully Recovered from end of procedure
Time to Fully Alert from end of procedure
Change from baseline DSST score over time during recovery period
Modified OAA/S scores over time during the dosing initiation, procedural, and recovery periods
Duration and percent of time when a patient's Modified OAA/S score is at each level between the first dose of study medications and Fully Alert, inclusive
Duration of sedation
Number of doses of study medication administered for the procedure
Time to sedation
Number of procedure interruptions due to inadequate sedation
Patient's rating of experience after Fully Recovered
Patient's rating at 24 hour post-discharge telephone survey
Investigator's rating at end of procedure
Blinded evaluator's rating after patient is Fully Recovered
Safety Endpoints
Nature, frequency, severity, relationship to treatment, and outcome of all adverse events
Sedation-related adverse events and interventions
Laboratory parameters and vital signs
Airway assistance
Concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD, PharmD, Study Director — Eisai Inc.